CLINICAL TRIAL: NCT03651089
Title: Safety, Tolerability and Pharmacokinetics of a Single Subcutaneous Administration of SP16-a SERPIN-like, Small Peptide Agonist of the Low Density Lipoprotein-like Receptor 1-in Healthy Individuals
Brief Title: SP16 SERPIN-like Peptide Administration in Healthy Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serpin Pharma, LLC (Other)
Collaborators: George Mason University (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-SP16
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Participants
Keywords: acute myocardial infarction; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This study is set up as 3 sequential parallel studies, each testing a different drug dosage against placebo. In each dosing cohort, three patients (2 active and 1 placebo) will be randomized to receive a single study drug infusion on separate days, at least 24 hours apart. The remaining subjects in each dosing cohort (1 placebo and 4 active) will receive study drug after at least 24 hours from the 3rd subject.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SP16 0.0125 (Active Comparator): 0.0125 mg/kg of SP16 will be administered by subcutaneous injection once
  Interventions: Drug: SP16
- SP16 0.050 (Active Comparator): 0.050 mg/kg of SP16 will be administered by subcutaneous injection once
  Interventions: Drug: SP16
- SP16 0.20 (Active Comparator): 0.20 mg/kg of SP16 will be administered by subcutaneous injection once
  Interventions: Drug: SP16
- placebo (Placebo Comparator): Placebo (sterile saline) will be administered by subcutaneous injection once
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: SP16 — subcutaneous injection of experimental anti-inflammatory drug
  Arms: SP16 0.0125; SP16 0.050; SP16 0.20
Drug: Placebos — subcutaneous injection of sterile saline
  Arms: placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled Phase 1 Clinical Trial of 24 healthy individuals to test the safety, tolerability and pharmacokinetics of a single subcutaneous administration of Serpin Peptide 16 (SP16), a Serine Protease Inhibitor (Serpin)-like, small peptide agonist of the Low Density Lipoprotein Receptor-like Protein 1 (LRPP1) hypothesized to have anti-inflammatory activity.

DETAILED DESCRIPTION:
One of the major determinants for outcome in patients with acute myocardial infarction (AMI) is the degree of inflammatory response. SP16 is a synthetic anti-inflammatory peptide developed to reproduce the anti-inflammatory activities of naturally occurring Serpins and has been tested as a treatment for AMI in mice. This Phase I trial will be the first to test the hypothesis that a single subcutaneous administration of SP16 is safe and well tolerated in healthy individuals, while also assessing the pharmacokinetic parameters of three different dosages. Participants will undergo direct clinical monitoring for up to 12 hours after drug administration. Additionally, participants will follow up with the same assessments at 24 hours, 48-72 hours and 7 days post drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 to 59 years
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability to take oral medication and be willing to adhere to the medication regimen
* For females of reproductive potential: Use of highly effective contraception
* For males of reproductive potential: Use of condoms

Exclusion Criteria:

* Acute or chronic illness affecting organ function or requiring medications (including, but not limited to, cardiovascular, hepatic, renal hematologic, neurologic, dermatologic, psychiatric, or rheumatologic disease);
* Febrile illness within the previous 14 days;
* Known allergic reactions to components of the study agent;
* Treatment with another investigational drug or other intervention within 30 days;
* Current tobacco use or tobacco use within 60 days;
* Household contacts who are immunocompromised;
* Chronic infection(s) (of any kind);
* Malignancy (of any kind);
* Substance abuse disorder(s);
* Pregnancy or breastfeeding;
* Any other conditions that would place the subject at increased risk of adverse events or interfere with the conduct or interpretation of the study, in the opinion of the investigators.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Preliminary Safety Assessment: Occurence of adverse events | 7 days follow-up
  Occurence of adverse events

SECONDARY OUTCOMES:
Volume of distribution of SP16 in healthy subjects | 7 days
  Population estimate of volume of distribution will be calculated using non-compartmental analysis
Clearance of SP16 in healthy subjects | 7 days
  Population estimate of clearance will be calculated using non-compartmental analysis

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to present the data promptly upon analysis as an abstract to a national meeting and/or manuscript

REFERENCES:
- See also: A phase 1 clinical trial of SP16, a first-in-class anti-inflammatory LRP1 agonist, in healthy volunteers — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0247357